CLINICAL TRIAL: NCT00249106
Title: Randomized, Placebo-Controlled, Dose-Escalating, Double-Blinded Phase 1 Safety and Immunogenicity Study of Clade C DNA Vaccine ADVAX e/g + ADVAX p/N-t (ADVAX) Administered Intramuscularly to HIV-Uninfected, Healthy Volunteers.
Brief Title: Safety and Immunogenicity of a Plasmid HIV Vaccine in HIV Uninfected Adults
Acronym: C001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Collaborators: Aaron Diamond AIDS Research Center (Other); University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IAVI C001
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2011-09

CONDITIONS: HIV Infection
MeSH Terms: conditions — HIV Infections | interventions — delta inulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HIV vaccine (Experimental): dosage escalation of ADVAX
  Interventions: Biological: ADVAX
- Placebo (Placebo Comparator): Sodium phosphate
  Interventions: Biological: ADVAX

INTERVENTIONS:
Biological: ADVAX
  Other Names: DNA HIV vaccine

SUMMARY:
The purpose of this study is to determine the safety and immune response to a investigational DNA Plasmid HIV vaccine, ADVAX e/g + ADVAX p/n-t (ADVAX), at three different dosage levels, in adults who are not infected with HIV.

DETAILED DESCRIPTION:
This is a dose escalation trial. Study site staff and volunteers will be blinded, blinding will not apply to the assignment of dose levels (low, middle or high).

Volunteers will be screened up to 42 days before vaccination and will be followed for 18 months after the first vaccination.

15 volunteers will be randomized in a 4:1 ratio of active vaccine to placebo. Safety and tolerability of the ADVAX e/g + ADVAX p/n-t investigational product will be evaluated at least 14 days after the tenth volunteer in the lower dosage group receives the second injection before proceeding to the nextdosage group.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult males and females;
* Age at least 18 years on the day of screening and no greater than 60 years on the day of the first vaccination;
* Available for follow up for the planned duration of the study (screening plus 18 months);
* In the opinion of the principal investigator or designee, has understood the information provided. Written informed consent needs to be given before any study-related procedures are performed;
* Willing to undergo HIV testing and counseling, and receive HIV test results;
* If sexually active female, using an effective method of contraception from screening until at least 4 months after last vaccination, and willing to undergo urine pregnancy test.
* If sexually active male, willing to use an effective method of contraception from screening until 4 months after the last vaccination.

Exclusion Criteria:

* Clinically relevant abnormality on history or examination including history of immunodeficiency or use of systemic corticosteroids, immunosuppressive, antiviral, anticancer, or other medications considered significant by the designated trial physician in last 6 months;
* Any acute or chronic medical condition requiring care of a physician (e.g.,, diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that, in the opinion of the investigator, would preclude participation;
* Any of the following abnormal laboratory parameters that are moderate, severe, or very severe: haematology (hemoglobin, absolute neutrophil count, absolute lymphocyte count, absolute CD4/CD8 count, platelets); urinalysis, biochemistries (total bilirubin, creatinine, AST, ALT). Volunteers with mild laboratory abnormalities that are judged by the principal investigator or designee to be not clinically significant may be enrolled.
* Reported high- risk behaviour for HIV infection, defined as:
* Had unprotected vaginal or anal sex with a known HIV infected person or a casual partner (i.e., no continuing established relationship) within 6 months before vaccination
* Engaged in sex work for money or drugs within 6 months before vaccination
* Used injection drugs (illicit), or Acquired an STD within 6 months before vaccination ;
* If female, pregnant or planning a pregnancy within 4 months after last vaccination or lactating;
* Receipt of blood transfusion or blood products 6 months prior to vaccination;
* Receipt of a live attenuated vaccine (other than influenza) within 30 days or other vaccine within 14 days of vaccination;
* Participation in another clinical trial of an investigational product currently or within past 12 weeks or expected participation during this study;
* Receipt of another experimental HIV vaccine at any time;
* Infected with HIV-1 or HIV-2 as indicated by ELISA and/or RT-PCR;
* History of severe local or systemic reaction to vaccination or history of severe allergic reactions;
* Confirmed diagnosis of hepatitis B (surface antigen, HbsAg); hepatitis C (HCV antibodies) or active syphillis;
* History of grand-mal epilepsy, or currently taking anti-epileptics;
* In the opinion of the investigator, unlikely to comply with protocol.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2003-12; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Safety of ADVAX | 18 months
  dose escalation study

SECONDARY OUTCOMES:
Immunogenicity of ADVAX | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: David Ho, MD, Principal Investigator — Aaron Diamond AIDS Research Center; Michael Keefer, MD, Principal Investigator — University of Rochester; Soe Than, MD, Study Director — International AIDS Vaccine Initiative
Locations (2):
- United States (2):
  - Rockefeller University Hospital, New York, New York
  - University of Rochester Medical Center, Rochester, New York

REFERENCES:
- [Result] Vasan S, Schlesinger SJ, Huang Y, Hurley A, Lombardo A, Chen Z, Than S, Adesanya P, Bunce C, Boaz M, Boyle R, Sayeed E, Clark L, Dugin D, Schmidt C, Song Y, Seamons L, Dally L, Ho M, Smith C, Markowitz M, Cox J, Gill DK, Gilmour J, Keefer MC, Fast P, Ho DD. Phase 1 safety and immunogenicity evaluation of ADVAX, a multigenic, DNA-based clade C/B' HIV-1 candidate vaccine. PLoS One. 2010 Jan 25;5(1):e8617. doi: 10.1371/journal.pone.0008617. PMID 20111582